CLINICAL TRIAL: NCT05223985
Title: EPISEEG - EPC Performance Investigation for StereoElectroEncephaloGraphy
Brief Title: EPC Performance Investigation for StereoElectroEncephaloGraphy
Acronym: EPISEEG
Status: Recruiting | Type: Observational
Sponsor: Alcis (Industry)
Responsible Party: Sponsor
Other Study IDs: EPISEEG
Record Dates: First submitted 2021-12-23; First posted 2022-02-04 (Actual); Last update posted 2024-08-05 (Actual); Status verified 2024-08

CONDITIONS: Epilepsy
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Depth Coagulation Electrode — SEEG and thermocoagulation

SUMMARY:
The objective of this multicentre study is to collect preoperative, intra operative, early, short, intermediate and mid-term(one years) on the related clinical complications and functional outcomes of market-approved Alcis products to demonstrate safety and performance of these devices in a real-world setting.

DETAILED DESCRIPTION:
Outcome data collected from this study will provide the basis for Post-Market Surveillance (PMS) reporting, Clinical Study Report (CSR), Clinical Evaluation Report (CER) on Alcis devices and support peer-reviewed publications on products performance and safety.

ELIGIBILITY:
Inclusion Criteria:

* To be included, patients must be:
* 18 months to 65 years
* Patient with drug-resistant and disabling focal epilepsy
* Informed and willing to sign an informed consent form approved by EC / For minors: if one of the parents cannot consent within the timeframe provided by the protocol, then only one parent's signature is required
* Affiliation to the social security or foreign regime recognized in France
* For prospective inclusion: Patient considered for SEEG exploration as part of pre-surgical assessment of epilepsy
* For ambispective inclusion:

  * Must have undergone an SEEG exploration with one ALCIS device before the date of the initiation visit
  * Follow-up visits (at least 12-month) must be prospective
  * Must have complete information available for each completed visit (demographics, preoperative information, implantation information, device details) *.

Exclusion Criteria:

* • Not able to comply with the study procedures based on the judgment of the assessor (e.g. cannot comprehend study questions, inability to keep scheduled assessment times)

  * Any medical condition that could impact the study at investigator's discretion (e.g. allergy…)
  * Pregnant women (contraindication to SEEG exploration)
  * Adult subject to legal protection measure
  * Skull thickness inferior at 2 mm

Ages: 18 Months to 65 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: The patient treated by Depth Coagulation Electrode is drug-resistant epilepsies patient.
Sampling Method: Probability Sample
Enrollment: 74 (Estimated)
Dates: Start 2022-04-29 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Signal quality | through study completion, an average of 10 days".
  percentage of contacts that measured a signal
Modification of Electroencephalography trace post-coagulation | through study completion, an average of 1 hours".
  Modification of Electroencephalography trace post-coagulation

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Centre d'Investigation Clinique : Equipe Timone Adultes CPCET, Marseille
  - Pôle Investigation - Fondation Adolphe de Rothschild, Paris, Île-de-France Region